CLINICAL TRIAL: NCT01528553
Title: Stapling Versus 8plate for Correction of Genu Valgus. A Randomised Clinical Study
Brief Title: Stapling Versus 8plate for Correction of Genu Valgus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VEK 20080179
Record Dates: First submitted 2012-01-20; First posted 2012-02-08 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Deformity; Genu Valgus
Keywords: genu valgus; lower limb; paediatric; epiphysiodesis
MeSH Terms: conditions — Congenital Abnormalities; Genu Valgum | interventions — Sutures

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Staples (Active Comparator): Old implant type
  Interventions: Device: Staples (Richards, Smith & Nephew)
- 8plate (Active Comparator): New implant type
  Interventions: Device: 8plate

INTERVENTIONS:
Device: 8plate — 12 mm or 16 mm plate. 24 mm or 36 mm screw
  Other Names: 8plate system
  Arms: 8plate
Device: Staples (Richards, Smith & Nephew) — Staples (3 on each side)
  Other Names: Richards staples, Smith & Nephew
  Arms: Staples

SUMMARY:
In children with excessive knock knees it may be necessary to use guided growth (small surgical procedure) so the child outgrows the condition before maturity. A new implant is on the market and the investigators compare this implant (8plate) with the old technique (staples) in a randomised setup.

The hypothesis is that the 8plate provides a faster correction rate and that this treatment is superior to stapling.

DETAILED DESCRIPTION:
Correcting angulating deformities of the lower limb is a subject of major interest in paediatric orthopaedics. Epiphysiodesis is the technique by which unilateral bone growth is stopped. Traditionally this has been performed with staple technique. The 8-plate technique is new and advocated because it is believed to reduce the risk of premature closure of the growth plate compared to stapling. The benefit of the 8-plate technique has not yet been proven in experimental or randomised clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic genu valgus
* At least one year of remaining growth

Exclusion Criteria:

* Unilateral conditions

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2009-08; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Treatment time | up to 104 weeks
  Will be followed with repeated clinical examinations until correction of deformity.

SECONDARY OUTCOMES:
Radiological correction | up to 104 weeks
  After correction of deformity.

CONTACTS AND LOCATIONS:
Overall Officials: Bjarne Møller-Madsen, Professor, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Background] Stevens PM. Guided growth for angular correction: a preliminary series using a tension band plate. J Pediatr Orthop. 2007 Apr-May;27(3):253-9. doi: 10.1097/BPO.0b013e31803433a1. PMID 17414005
- [Background] Jelinek EM, Bittersohl B, Martiny F, Scharfstadt A, Krauspe R, Westhoff B. The 8-plate versus physeal stapling for temporary hemiepiphyseodesis correcting genu valgum and genu varum: a retrospective analysis of thirty five patients. Int Orthop. 2012 Mar;36(3):599-605. doi: 10.1007/s00264-011-1369-5. Epub 2011 Oct 9. PMID 21983939
- See also: Research Group Page — http://dpor.dk/
- See also: Hospital Webpage — http://www.auh.dk/